CLINICAL TRIAL: NCT01416740
Title: A Prospective Comparison of Indirect and Direct MR Arthrography of the Shoulder Using Arthroscopic Correlation
Brief Title: A Comparison of Indirect and Direct MR Arthrography of the Shoulder Using Arthroscopic Correlation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty with recruitment, PI left the institution
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Robert Lyons M.D., Assistant Professor of Orthopaedic Surgery, Penn State Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 31905
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2011-08

CONDITIONS: Shoulder Pain
Keywords: Indirect magnetic resonance arthrogram; Direct magnetic resonance arthrogram; Diagnostic tests for shoulder pain
MeSH Terms: conditions — Shoulder Pain | interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indirect MRA (Experimental): After patient has signed consent and had blood tests to ensure normal kidney function (BUN and Creatinine) as well as serum and urine pregnancy tests for females to ensure there is no pregnancy, the patient will have an Indirect MRA. The participant will be weighed and the correct dose of 0.1 mmol/kg calculated. An IV will be inserted into participant's arm. The gadopentetate dimeglumine will be injected into the IV and the patient will be asked to gently exercise the shoulder (small windmills and flexion/extension) for 5 minutes. The patients then undergo MRI imaging 15-30 minutes after the injection. Contraindications include known allergy to gadopentetate dimeglumine, and renal failure with creatinine clearance of less than 30ml/min.
  Interventions: Procedure: Indirect MRA of shoulder; Drug: Gadopentetate Dimeglumine

INTERVENTIONS:
Procedure: Indirect MRA of shoulder — Patient will be weighed and the correct dose of 0.1 mmol/kg calculated. An IV will be inserted into patient's arm. The gadopentetate dimeglumine will be injected into the IV and the patient is asked to gently exercise the shoulder (small windmills and flexion/extension) for 5 minutes. The patients then undergo MRI imaging 15-30 minutes after the injection. Contraindications include known allergy to gadopentetate dimeglumine, and renal failure with creatinine clearance of less than 30ml/min.
Drug: Gadopentetate Dimeglumine — Patient will be weighed and the correct dose of 0.1 mmol/kg calculated. An IV will be inserted into patient's arm. The gadopentetate dimeglumine will be injected into the IV and the patient is asked to gently exercise the shoulder (small windmills and flexion/extension) for 5 minutes. The patients then undergo MRI imaging 15-30 minutes after the injection. Contraindications include known allergy to gadopentetate dimeglumine, and renal failure with creatinine clearance of less than 30ml/min.
  Other Names: gadolinium DTPA; Magnevist

SUMMARY:
This study will prospectively compare the findings of two diagnostic tests, Direct Magnetic Resonance Arthrography(MRA) and Indirect MRA, to the findings during shoulder arthroscopy in patients with shoulder pain. The sensitivity and specificity of both Direct and Indirect MRA's in diagnosing specific pathologies of the shoulder will be determined using shoulder arthroscopy as the gold standard.

DETAILED DESCRIPTION:
Direct MR arthrography (MRA) requires the injection of a contrast agent into the shoulder under fluoroscopic or ultrasound guidance, followed by magnetic resonance imaging (MRI). This is invasive, risks infection, and requires time and resources. It has recently been shown that the intravenous administration of gadopentetate dimeglumine enhances the joint cavity during an MRI and thus indirectly produces an arthrographic effect(Indirect MRA). The study will enroll patients who have already had a Direct MRA as part of their standard of care diagnostic test for shoulder pain, if it is determined by their surgeon that arthroscopic surgery is indicated they will be asked if they would be willing to have an Indirect MRA prior to their arthroscopic surgery. The patient will need to have a blood test(BUN and Creatinine)done to ensure kidney function is normal, and a serum and urine pregnancy test, if female, to ensure there is no pregnancy, prior to the completion of the Indirect MRA. After the patient's scheduled shoulder arthroscopic surgery, the results of the two MR arthrography techniques will be compared for sensitivity and specificity in detecting partial and full thickness rotator cuff tears, labral tears, long head biceps dislocation/tearing, and grade IV cartilage lesions by comparing the results to the actual arthroscopic findings. The Direct MR arthrography and arthroscopic surgery are standard of care and would occur regardless of this study, the Indirect MR arthrography is the diagnostic intervention that is study-related.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 - 70 years old
* Continued shoulder pain for 2 months duration that limits his/her activity despite conservative treatment
* Had a standard of care Direct MR arthrogram performed from which the surgeon determined that arthroscopic surgery was indicated.

Exclusion Criteria:

Clinical Evidence of

* Tumor
* Infection
* Previous shoulder surgery
* Contraindication for MRI
* Allergy to contrast
* Coagulopathy
* Known allergy to gadolinium DTPA
* Renal failure with creatinine clearance of less than 30ml/min
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of Direct and Indirect MR Arthrograms in detecting pathologies of the shoulder when compared with Arthroscopic findings. | Patients will be foollowed from their Indirect MRA to their arthoscopic shoulder surgery, approximately one month from time of consent
  This study will compare the findings of the Indirect MRA and the retrospective data of the Direct MRA, to the results obtained during their arthroscopic shoulder surgery in patients with shoulder pain. The incidence of partial and full thickness rotator cuff tears, long head biceps dislocation/tearing, and grade IV cartilage lesions will be recorded for each type of MRA of the shoulder. The sensitivity and specificity of both direct and indirect MR arthrography in diagnosing shoulder problems will be determined by what was actually visualized during their arthroscopic shoulder surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lyons, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Bone and Joint Institute, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Jung JY, Yoon YC, Yi SK, Yoo J, Choe BK. Comparison study of indirect MR arthrography and direct MR arthrography of the shoulder. Skeletal Radiol. 2009 Jul;38(7):659-67. doi: 10.1007/s00256-009-0660-7. Epub 2009 Feb 19. PMID 19225775
- [Background] Oh DK, Yoon YC, Kwon JW, Choi SH, Jung JY, Bae S, Yoo J. Comparison of indirect isotropic MR arthrography and conventional MR arthrography of labral lesions and rotator cuff tears: a prospective study. AJR Am J Roentgenol. 2009 Feb;192(2):473-9. doi: 10.2214/AJR.08.1223. PMID 19155413
- [Background] Herold T, Bachthaler M, Hamer OW, Hente R, Feuerbach S, Fellner C, Strotzer M, Lenhart M, Paetzel C. Indirect MR arthrography of the shoulder: use of abduction and external rotation to detect full- and partial-thickness tears of the supraspinatus tendon. Radiology. 2006 Jul;240(1):152-60. doi: 10.1148/radiol.2393050453. Epub 2006 May 18. PMID 16709790
- [Background] Dinauer PA, Flemming DJ, Murphy KP, Doukas WC. Diagnosis of superior labral lesions: comparison of noncontrast MRI with indirect MR arthrography in unexercised shoulders. Skeletal Radiol. 2007 Mar;36(3):195-202. doi: 10.1007/s00256-006-0237-7. Epub 2006 Dec 1. PMID 17139503